CLINICAL TRIAL: NCT06836531
Title: POCT Detection for Blood Concentration of Tirofiban in Acute Myocardial Infarction Based on Azo-POP Probe, and Use Metabolomics Analysis Combined with Machine Learning Algorithms for Screening Biomarkers of Myocardial Infarction.
Brief Title: POCT Detection for Blood Concentration of Tirofiban in Acute Myocardial Infarction Based on Azo-POP Probe.
Status: Enrolling by invitation | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Other Study IDs: 2024135A; 2023S193 (Other Grant/Funding Number: Ningbo Public Welfare Research Program)
Record Dates: First submitted 2024-11-28; First posted 2025-02-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy: those without coronary atherosclerotic heart disease
- AMI: those with acute myocardial infarction but without percutaneous coronary intervention
- AMI-PCI: those with acute myocardial infarction and percutaneous coronary intervention

SUMMARY:
The goal of this observational study is to monitor blood drug concentration during the use of tirofiban, predict the occurrence of intraoperative and postoperative complications related to interventional therapy, and evaluate the efficacy of multiple antiplatelet drugs.The main question it aims to answer is:

1. If the POCT detection technology for blood concentration of tirofiban based on portable mass spectrometer can be used for on-site sampling, clinical testing, and immediate analysis next to patients undergoing coronary intervention therapy.
2. LC-MS/MS untargeted metabolomics analysis techniques combined with machine learning algorithms will be used to screen biomarkers for myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* The patient meets the diagnostic criteria for STEMI (refer to the "Diagnosis and Treatment Guidelines for Acute ST Segment Elevation Myocardial Infarction (2019)")
* The onset time is less than 12 hours
* Agree to perform direct PCI
* Heart function (Killip class) ≤ Level III
* There are no direct PCI contraindications.

Exclusion Criteria:

* Patients allergic to tirofiban or/and aspirin
* Patients with a history of intracranial hemorrhage
* Patients with stroke/transient ischemic attack within six months
* Patients who have taken oral anticoagulants within 30 days before admission and cannot stop taking them
* Patients receiving clopidogrel or ticagrelor from other manufacturers or formulations due to directive events
* Patients who have received or plan to undergo fibrinolysis therapy within 24 hours
* Patients with a history of major surgery within 30 days, or those who plan to undergo major surgery during the study process
* Patients with a history of gastrointestinal bleeding within 6 months, or those with severe bleeding disorders or tendencies towards bleeding
* Patients with severe combined liver and kidney dysfunction
* Refuse to participate in this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are diagnosed with acute myocardial infarction and treated with direct PCI in the cardiology department of our hospital during the project execution period.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Establish a POCT detection technology for blood concentration of tirofiban based on portable mass spectrometer, which can perform on-site sampling, clinical testing, and immediate analysis during PCI. | From enrollment to the end of treatment at 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No